CLINICAL TRIAL: NCT03078725
Title: Failure Rate of GLyburide And Metformin Among Gestational Diabetics
Acronym: GLAM
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Research was competing with other projects in the department, and no patients were recruited.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Jenifer Dinis Ballestas, Medical Doctor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-16-1052
Record Dates: First submitted 2017-03-07; First posted 2017-03-13 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Gestational Diabetes Mellitus, Class A2
Keywords: gestational diabetes; glyburide; metformin; failure rate
MeSH Terms: conditions — Diabetes, Gestational | interventions — Glyburide; Metformin

STUDY DESIGN:
Intervention Model Description: patients will be randomized to two groups, one receiving glyburide and one receiving metformin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Glyburide (Active Comparator): hypoglycemic agent approved for treatment of GDMA2
  Interventions: Drug: Glyburide
- Metformin (Active Comparator): hypoglycemic agent approved for treatment of GDMA2
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Glyburide — oral hypoglycemic agent
  Arms: Glyburide
Drug: Metformin — oral hypoglycemic agent
  Arms: Metformin

SUMMARY:
A pragmatic, comparative effectiveness trial of glyburide versus metformin.

DETAILED DESCRIPTION:
Patients with gestational diabetes requiring pharmaceutical treatment will be randomized to receive glyburide or metformin. Dose increases will be determined by the patient's physician. Patients will be determined to have failed either medication if glucose control can not be achieved with the maximum dose of the medication, if insulin is stared to achieve glucose control or if another oral agent is started along for glucose control.

ELIGIBILITY:
Inclusion Criteria:

We will include women between 20 and 34 weeks gestational age, with a diagnosis of GDM as per the following criteria:

* 1 hour Glucose tolerance test of >130 mg/dl, followed by two abnormal values on 3 hour Glucose tolerance test, or:
* A single 1 hour Glucose tolerance test value of > 200 mg/dl, and:
* Failure to achieve glycemic control with diet and exercise or deemed to require pharmacological therapy as per physician's criteria

Exclusion Criteria:

* - Known renal impairment.
* Known hepatic disease.
* Pre-gestational diabetes.
* Known allergy to glyburide, metformin or sulfa drugs.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06-20 (Estimated); Primary Completion 2018-03-10 (Estimated); Study Completion 2018-05-10 (Estimated)

PRIMARY OUTCOMES:
Failure rate | from onset of oral therapy until delivery
  need to start insulin therapy or another hypoglycemic agent during the pregnancy to maintain normal glucose levels or need for delivery due to hyperglycemia.

SECONDARY OUTCOMES:
Mean overall plasma glucose | from enrollment to delivery
  average of all postprandial glucose measurements
Mean weekly fasting glucose | from enrollment to delivery
  average of all fasting glucose measurements
preeclampsia | from enrollment to delivery
  preeclampsia
cesarean section | from enrollment to delivery
  mode of delivery
neonatal hypoglycemia | from enrollment to delivery
  neonatal hypoglycemia
LGA infant | from enrollment to delivery
  LGA infant
birthweight > 4500 grams | from enrollment to deliveryfrom enrollment to delivery
  birthweight > 4500 grams
gestational age at birth | from enrollment to delivery
  gestational age at birth
incidence of medication side effects | from enrollment to delivery
  nausea, emesis, diarrhea, abdomainal bloating

IPD SHARING:
Plan to Share IPD: No